CLINICAL TRIAL: NCT05320835
Title: A Geospatial Analysis of Hotspots and Targeted Injection Settings Pilot Intervention for HIV Prevention Among People Who Inject Drugs in Baltimore, Maryland
Brief Title: A Setting Focus Overdose Prevention Intervention
Acronym: Oasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01DA050470 (NIH); IRB00019139 (Other: JHSPH IRB); R01DA050470 (NIH)
Record Dates: First submitted 2022-03-30; First posted 2022-04-11 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; HCV; Drug Overdose
MeSH Terms: conditions — HIV Infections; Drug Overdose | interventions — Seroconversion

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial (RCT)
Who Masked: Participant
Masking Description: Equal attention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): behavioral training with 6 sessions
  Interventions: Behavioral: HIV, HCV and overdose prevention
- comparison (Active Comparator): Attention control
  Interventions: Behavioral: HIV, HCV and overdose prevention

INTERVENTIONS:
Behavioral: HIV, HCV and overdose prevention — HIV, HCV and overdose prevention

SUMMARY:
A pilot injection-setting targeted peer-driven intervention to reduce HIV and hepatitis C virus transmission and overdose risk behaviors among people who inject drugs (PWID).

DETAILED DESCRIPTION:
This is a pilot of an injection setting targeted peer-driven intervention to reduce HIV/HCV transmission and overdose risk behaviors. Participants will be randomized to conditions: 1) Peer education and stocking of semi-public injection settings (SPIS) with risk reduction materials, and the standard of care. Based on their SPIS use, 120 index PWID participants will be selected.

A conceptual model for the intervention: The conceptual model is based on social influence, social network, and social cognitive theory. The prior work delineated social influence mechanisms. It is expected that training and modeling of effective communication skills will increase the occurrence of conversations on HIV/HCV and overdose prevention. These conversations will then alter perceived descriptive and prescriptive social norms of risk behaviors. The prior work is being enhanced by increasing the availability of risk reduction materials as well as the cuing and modeling risk reduction behaviors in risk settings. It has been found that PWID are motivated to conduct peer education; it enhances their status and provides them a prosocial role in the community. It is hypothesized that peer outreach and supply of materials to SPIS will lead to reduced sharing of injection equipment and increased naloxone availability.

ELIGIBILITY:
Inclusion Criteria:

* Current drug user (opioid use in the prior two weeks)

Exclusion Criteria:

* Any mental or physical health impairment that impedes ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Overdose prevention | 6 months
  Frequency of carrying naloxone
HIV/HCV prevention | 6 months
  Frequency of using used cookers

SECONDARY OUTCOMES:
Overdose behaviors | 6 months
  Frequency of testing drugs before using
Overdose behaviors 2 | 6 months
  Frequency of talking about overdose prevention

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Lighthouse Studies at Peer Point, Baltimore, Maryland, United States